CLINICAL TRIAL: NCT07290244
Title: A Phase 1 Single Dose Study to Evaluate the Safety and Tolerability of ER-100 in Optic Neuropathies [Open Angle Glaucoma (OAG) and Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)]
Brief Title: Evaluating ER-100 for Safety in People With Glaucoma or Non-Arteritic Anterior Ischemic Optic Neuropathy (Optic Nerve Conditions)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Life Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB100-001
Record Dates: First submitted 2025-11-19; First posted 2025-12-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Open Angle Glaucoma (OAG); NAION( Non-arteritic Anterior Ischemic Optic Neuropathy)
Keywords: Optic Neuropathy; Retinal Diseases; Aging/Cellular Aging; Open-Angle Glaucoma; Non-Arteritic Anterior Ischemic Optic Neuropathy; Partial Epigenetic Reprogramming; Epigenetic Therapy
MeSH Terms: conditions — Glaucoma, Open-Angle; Optic Nerve Diseases; Retinal Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a sequential cohort design. Participants with Open Angle Glaucoma (OAG) are enrolled first in a dose escalation phase to evaluate safety and tolerability at multiple dose levels. Each dose level begins with a sentinel participant followed by additional participants after Safety Review Committee (SRC) evaluation. Upon completion of the OAG cohort, a dose is selected for the Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION) cohort. NAION participants are enrolled in a dose expansion phase, beginning with limited enrollment and SRC review prior to cohort expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OAG - Low Dose ER-100 (2 x 10^11 vg/eye) (Experimental): Participants with Open Angle Glaucoma will receive a low dose of ER-100 administered to one eye. ER-100 is delivered via a modified adeno-associated virus (AAV) vector and activated by systemic doxycycline taken for 8 weeks (56 days). This dose level begins with a sentinel participant followed by additional participants after SRC review.
  Interventions: Genetic: ER-100 epigenetic therapy
- OAG - High Dose ER-100 (6 x 10^11 vg/eye) (Experimental): Participants with Open Angle Glaucoma will receive a higher dose of ER-100 administered to one eye. ER-100 is delivered via a modified AAV vector and activated by systemic doxycycline for 8 weeks. This dose level also begins with a sentinel participant and proceeds following SRC review.
  Interventions: Genetic: ER-100 epigenetic therapy
- NAION - Selected Dose ER-100 (Experimental): Participants with Non-Arteritic Anterior Ischemic Optic Neuropathy will receive ER-100 at a dose selected based on safety and tolerability data from the OAG cohort. ER-100 is administered to one eye and activated by systemic doxycycline for 8 weeks. Initial enrollment is limited to three participants, with potential expansion to six following SRC review.
  Interventions: Genetic: ER-100 epigenetic therapy

INTERVENTIONS:
Genetic: ER-100 epigenetic therapy — ER-100 is an investigational AAV-based epigenetic therapy administered via intravitreal injection to one eye. It uses a modified adeno-associated virus (AAV) vector to deliver instructions for producing three transcription factors-OCT4, SOX2, and KLF4 (collectively referred to as OSK)-intended to reverse age-related epigenetic changes in retinal cells. Systemic doxycycline is administered for 8 weeks (56 days) to activate OSK expression. ER-100 does not alter the participant's existing genes, and the AAV vector has been engineered to eliminate its ability to cause infectious disease.
  Other Names: OSK epigenetic therapy; Investigational epigenetic therapy for optic neuropathies

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of a single dose of ER-100 in adults with optic nerve conditions, specifically Open Angle Glaucoma (OAG) and Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION). The main questions it aims to answer are:

* Is ER-100 safe when given as a single dose to people with OAG or NAION
* What side effects may occur, if any, after taking ER-100?

Participants will:

* Receive a single dose of ER-100
* Undergo safety assessments including detailed eye examination and laboratory tests
* Provide body fluid samples (tears, saliva, feces, urine) to help researchers understand how the drug is processed and cleared from the body
* Complete questionnaires about their quality of life
* Be followed for up to 5 years to monitor long-term health and vision outcomes

DETAILED DESCRIPTION:
This first-in-human (FIH), Phase 1 clinical trial is designed to evaluate the safety and tolerability of ER-100, an investigational epigenetic therapy candidate intended for age-related optic neuropathies, such as Open Angle Glaucoma (OAG) and Non Arteritic Anterior Ischemic Optic Neuropathy(NAION) Over time, factors such as age, disease, injury, and lifestyle can leave marks on cells that affect how genes function. These marks, known as epigenetic changes, may contribute to cellular decline. ER-100 is designed to address cellular aging through epigenetic reprogramming. It works by delivering genetic instructions for producing three proteins-collectively referred to as OSK-that may help reverse these changes and restore cells to a more youthful state.

The therapy deployed in this trial uses a modified adeno-associated virus (AAV) vector to deliver OSK to retinal cells. The AAV has been engineered to remove its ability to cause infectious disease. Systemic doxycycline is administered for 8 weeks (56 days) to activate OSK expression. ER-100 does not alter the participant's existing genes.

The study includes two sequential cohorts: a dose escalation phase in participants with OAG, followed by a dose expansion phase in participants with NAION. In OAG, optic nerve damage is caused by increased intraocular pressure; in NAION, it results from sudden loss of blood flow. Both conditions lead to retinal cell damage and vision loss. ER-100 is intended to reduce this damage by reprogramming affected cells, potentially preserving or restoring vision.

At least two dose levels will be evaluated in the OAG cohort. The first ("sentinel") participant at each new dose level will receive ER-100 and be monitored for 28 days with review of data by a Safety Review Committee (SRC) prior to granting administration of ER-100 to 2 additional participants at that dose level. Dose escalation/reduction will proceed for subsequent participants in accordance with safety data and oversight from the SRC.

Once the dose escalation in OAG is complete, a dose will be selected for NAION after a consultation between the SRC and Sponsor. Initially only up to 3 NAION participants will be enrolled at the selected dose. After at least one NAION participant has completed 28 days of follow-up, the SRC will review safety data. All participants' data available at that time will be provided to the SRC for the review. Upon recommendation from the SRC, NAION enrollment may then continue up to a total of 6 NAION participants.

Up to 18 participants are planned for enrollment: 12 with OAG and 6 with NAION. A total of 14 clinic visits is planned for the study: 9 in the first 6 months, then one visit per year through Year 5. Additionally, there will be approximately 3 remote (telephone) visits.

This study represents the first administration of ER-100 in humans, following preclinical evaluation in laboratory models.

In this study, results are compared to baseline, which refers to assessments and study procedures at the first study visit and prior to ER-100 administration.

ELIGIBILITY:
Inclusion Criteria:

* Have clear eye structures and be able to have your pupils safely dilated so the doctor can examine the back of your eye.
* Able to understand the study and sign a consent form.
* Be between 40 and 85 years old.
* Willing and able to follow the study schedule, including all visits and tests, and speak a language for which the study materials are available.
* If a participant can become pregnant, must agree to use a condom and one highly effective form of birth control during sex for at least 4 months after receiving the study drug (ER-100).

For participants with open-angle glaucoma (OAG):

* Diagnosis of open-angle glaucoma in the study eye.
* Eye pressure must be less than 30 mmHg, measured with a standard test.
* Visual field test must show moderate to advanced vision loss (MD score between -6 and -20 dB).
* Not expected to need glaucoma surgery in the study eye within 2 months after receiving ER-100.
* Have reasonably good vision in the study eye (at least 20/80 on a standard eye chart).

For participants with NAION (non-arteritic anterior ischemic optic neuropathy):

* Had a sudden, painless loss of vision in one eye within 14 days before receiving ER-100, confirmed by a specialist. Having had NAION in the other eye is okay.
* The affected eye must show swelling of the optic nerve.
* Visual field test must show vision loss consistent with optic nerve damage (MD worse than -3.0 dB).
* If only one eye is affected, there must be a difference in pupil response between the two eyes.
* Have vision in the affected eye between 20/40 and 2/500 on a standard eye chart.

Exclusion Criteria:

* History of optic neuritis (inflammation of the optic nerve) or repeated episodes of eye inflammation (uveitis) not caused by injury or surgery.
* Allergic reactions to tetracycline antibiotics or steroid medications.
* Moderate to severe cataracts, macular problems, or corneal issues that could interfere with eye testing.
* Unable to keep your eyes focused on a target during testing.
* Had cataract surgery or other eye surgery (including laser procedures) within 3 months before receiving the study drug.
* Had cancer (except for basal cell skin cancer) within the past 5 years.
* Have Type 1 diabetes, or poorly controlled Type 2 diabetes (A1c greater than 7 despite treatment).
* Have memory or thinking problems that prevent you from understanding the study or completing the required tests.
* Pregnant or breastfeeding.
* Have a weakened immune system, including a history of organ transplant, or test positive for HIV, hepatitis B or C, or tuberculosis.
* Have any other condition that, in the opinion of the study doctor, could increase your risk from the study drug or procedures, affect the study results, or make it hard for you to complete the study.
* Have macular disease, advanced diabetic eye disease, or other eye conditions that limit vision in the study eye.
* Eye pressure at screening is 30 mmHg or higher.
* Taking certain medications (warfarin, dilantin, carbamazepine, or barbiturates) within 14 days before starting the study or during the first 8 weeks.
* Have any other eye or vision problem that, in the opinion of the study doctor, could affect safety or interfere with vision testing.
* Have previously received any gene therapy using adeno-associated virus (AAV).

Additional Exclusion Criteria for Participants with Open-Angle Glaucoma (OAG):

- Diagnosed with glaucoma before age 40.

Additional Exclusion Criteria for Participants with NAION:

* Show signs of giant cell arteritis (a type of blood vessel inflammation), based on abnormal blood tests.
* Had NAION start in both eyes at the same time.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This outcome tracks any new or worsening health problems that occur while participants are receiving and completed oral doxycycline.
  These health problems are called treatment-emergent adverse events (TEAEs). Researchers record how often these events happen as well as their nature and seriousness.
  This helps determine whether ER-100 causes any short-term side effects during this phase.
Incidence of Dose-Limiting Toxicities During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This outcome measures how often participants experience dose-limiting toxicities, which are side effects serious enough to prevent increasing the dose, while receiving and completed oral doxycycline.
  These toxicities are defined by the study protocol and may differ for participants with open-angle glaucoma (OAG) and non-arteritic anterior ischemic optic neuropathy (NAION).
  This helps identify the highest dose that can be given safely during treatment.
Change in Safety Laboratory Tests (Liver Function Tests - LFTs) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Liver function tests (LFTs) measure specific enzymes and proteins in a blood sample to check how well the liver is working. These include alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), and lactate dehydrogenase (LDH). When liver cells are injured, these enzymes leak into the bloodstream, and higher levels on a blood test can signal a problem. Compared to baseline, higher levels can mean the liver is under stress or injured. Unit of Measure: Units per liter (U/L)
Change in Safety Laboratory Tests (Blood Protein Levels) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Blood proteins such as albumin and total protein help show nutritional status and how well the liver is making proteins. Compared to baseline, lower levels can mean poor nutrition or liver problems. Unit of Measure: Grams per deciliter (g/dL)
Change in Safety Laboratory Tests (Calcium, Glucose, Bilirubin, Creatinine, Blood Urea Nitrogen) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  These tests show how the body manages minerals, sugar, and waste. Calcium helps with bone and muscle function. Glucose shows blood sugar control. Bilirubin shows liver health. Creatinine and blood urea nitrogen (BUN) show kidney function. Compared to baseline, higher or lower levels can mean problems with the liver, kidneys, or metabolism. Unit of Measure: Milligrams per deciliter (mg/dL)
Change in Safety Laboratory Tests (Electrolytes: Sodium, Potassium, Chloride) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Electrolytes help keep the body's fluids and nerves working properly. Changes can mean dehydration or kidney problems. This outcome looks at how much sodium (Na), potassium (K), and chloride (Cl) levels change from baseline. Unit of Measure: Millimoles per liter (mmol/L)
Change in Safety Laboratory Tests (Electrolytes: Bicarbonate and Magnesium) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Bicarbonate helps control the body's acid balance. Magnesium is important for muscles and nerves. Changes can mean metabolic or kidney problems. This outcome looks at how much these levels change from baseline. Unit of Measure: Milliequivalents per liter (mEq/L)
Change in Safety Laboratory Tests (Hemoglobin) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Hemoglobin is a protein in red blood cells that carries oxygen. Lower levels can mean anemia, which is when the blood cannot carry enough oxygen. This outcome looks at how much hemoglobin changes from baseline. Unit of Measure: Grams per deciliter (g/dL)
Change in Safety Laboratory Tests (Hematocrit) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Hematocrit shows the percentage of blood made up of red blood cells. Compared to baseline, lower levels can mean anemia, which is when the blood cannot carry enough oxygen. Unit of Measure: Percent (%)
Change in Safety Laboratory Tests (White Blood Cell and Platelet Counts) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  White blood cells help fight infection. Platelets help blood clot. Compared to baseline, changes can mean infection, immune problems, or bleeding risk. Unit of Measure: Billion cells per liter (x10^9/L)
Change in Safety Laboratory Tests (Red Blood Cell Count) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Red blood cells carry oxygen throughout the body. Compared to baseline, lower levels can mean anemia, which is when the blood cannot carry enough oxygen. Unit of Measure: Trillion cells per liter (x10^12/L)
Change in Safety Laboratory Tests (Erythrocyte Sedimentation Rate) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This test shows inflammation in the body. Compared to baseline, higher values can mean infection or other inflammatory conditions. Unit of Measure: Millimeters per hour (mm/hr)
Change in Safety Laboratory Tests (C-Reactive Protein) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  C-reactive protein shows inflammation in the body. Compared to baseline, higher values can mean infection or other inflammatory conditions. Unit of Measure: Milligrams per liter (mg/L)
Change in Safety Laboratory Tests (Urine Test Results) During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  Urine tests check for blood, protein, sugar, and other substances. Compared to baseline, changes can mean kidney or urinary tract problems. Unit of Measure: Presence or absence
Change from Baseline in the Intraocular Pressure (IOP) in the Treated Eye During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures changes in pressure inside the treated eye while participants are receiving and completed oral doxycycline.
  Eye pressure is measured in millimeters of mercury (mmHg).
  On Day 1, pressure is measured using an instrument named Goldmann Applanation Tonometry (GAT), which is the gold standard. This instrument will gently touch the eye with a probe after applying numbing drops.
  After Day 1, pressure is measured using another, non-contact method, which uses a puff of air.
  If pressure increases significantly, GAT may be repeated to confirm.
  Depending on their values, higher or lower pressures compared to the participant's baseline may indicate safety concerns related to the treatment.
Change from Baseline in the Best Corrected Visual Acuity (BCVA) Letter Score in the Treated Eye During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in visual clarity (corrected with glasses or contact lenses for refractive errors like nearsightedness, farsightedness, or astigmatism) in the treated eye while participants are receiving and completed oral doxycycline.
  BCVA is assessed using a special chart called the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
  The number of letters read correctly is recorded as a letter score, ranging from 0 to 100. A drop in score from the baseline may indicate a safety issue affecting vision, while stable or improved scores suggest no adverse impact.
  Trial frames with the lens prescription determined at screening will be used for these assessments.
Change from Baseline in Humphrey Visual Field (HVF) Test Results During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in central and peripheral (side) field of vision while participants are receiving and completed oral doxycycline.
  The field of vision is assessed using the Humphrey Visual Field (HVF) test, which checks how well a person can see lights that flash in different areas of their visual field while they focus on a central point.
  Results are reported as a Mean Deviation (MD) score in decibels (dB). For participants with open-angle glaucoma (OAG), the test uses the SITA Standard 24-2 protocol. For participants with non-arteritic anterior ischemic optic neuropathy (NAION), a larger light stimulus (size V) is used.
  Compared to baseline, a more negative MD score means more vision loss, and a significant worsening in MD may suggest a safety concern.
Change from Baseline in Pattern Electroretinogram (pERG) During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in retinal function while participants are receiving and completed oral doxycycline.
  The pERG is a test that checks how well the retina responds to visual patterns like black and white stripes. It helps evaluate the health of retinal ganglion cells, which are important for sending visual signals to the brain.
  The test provides two types of results:
  * Amplitude (measured in microvolts, µV): This shows the strength of the retina's response.
  * Peak time (measured in milliseconds, ms): This shows how quickly the retina responds.
  Lower amplitudes or slower response times than those recorded at baseline may indicate worsening retinal function. A significant decline in these results may suggest a safety concern related to disease progression or if there are signs that the treatment is causing effects.
Change from Baseline in Quantitative Contrast Sensitivity Function (qCSF) During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in contrast sensitivity while participants are receiving and completed oral doxycycline.
  The quantitative Contrast Sensitivity Function (qCSF), also called quick CSF, is a computerized test that evaluates how well a person can detect differences in contrast, for example, the ability to discern subtle differences in shading or light and dark between an object and its background.
  Lower scores than those recorded at baseline may indicate worsening visual function, and a significant decline in one or more parameters may suggest a safety concern. Changes in these scores are monitored to detect potential trea
Change from Baseline in Optical Coherence Tomography (OCT): Ganglion Cell Layer (GCL) Thickness During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in the thickness of the ganglion cell layer (GCL) while participants are receiving and completed oral doxycycline.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using an instrument called the Heidelberg Spectralis system.
  The GCL contains the cell bodies of retinal ganglion cells, which are critical for transmitting visual information from the retina to the brain. GCL thickness is measured in micrometers (µm).
  A significant decrease in GCL thickness from baseline may suggest a safety concern related to disease progression or if there are signs that the treatment is causing effects.
Change from Baseline in Optical Coherence Tomography (OCT): Retinal Nerve Fiber Layer (RNFL) Thickness During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures the change in the thickness of the retinal nerve fiber layer (RNFL) while participants are receiving and completed oral doxycycline.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using the Heidelberg Spectralis system.
  The RNFL contains nerve fibers that help carry visual signals from the eye to the brain. RNFL thickness is measured in micrometers (µm).
  A significant decrease in RNFL thickness from baseline may suggest a safety concern related to disease progression or if there are signs that the treatment is causing effects.
Change from Baseline in Slit Lamp Exam Results During and Post-Doxycycline Activation Period - Safety | Baseline to Day 56, Day 112
  This outcome measures changes in the health of the front structures of the eye while participants are receiving and completed oral doxycycline.
  A slit lamp exam is a routine eye test that uses a bright light and microscope to closely examine the front parts of the eye, including the cornea, iris, lens, and the white part of the eye. The exam helps detect signs of irritation, inflammation, infection, or other possible damage.
  Changes from baseline observed during the slit lamp exam might be signs that the treatment is causing effects or that the disease is getting worse.

SECONDARY OUTCOMES:
Change from Baseline in the Intraocular Pressure (IOP) in the Treated Eye During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in pressure inside the treated eye while participants are receiving and completed oral doxycycline.
  Eye pressure is measured in millimeters of mercury (mmHg).
  On Day 1, pressure is measured using an instrument named Goldmann Applanation Tonometry (GAT), which is the gold standard. This instrument will gently touch the eye with a probe after applying numbing drops.
  After Day 1, pressure is measured using another, non-contact method, which uses a puff of air.
  If pressure increases significantly, GAT may be repeated to confirm.
  Lower pressures compared to baseline may indicate disease improvement.
Change from Baseline in the Intraocular Pressure (IOP) in the Treated Eye - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures changes in pressure inside the treated eye after participants stop taking oral doxycycline during the long-term follow-up period.
  Eye pressure is measured in millimeters of mercury (mmHg).
  On Day 1, pressure is measured using Goldmann Applanation Tonometry (GAT), which gently touches the eye with a probe after applying numbing drops.
  After Day 1, pressure is measured using non-contact tonometry, which uses a puff of air.
  If pressure increases significantly, GAT may be repeated to confirm.
  Depending on their values, higher or significantly lower pressures compared to the participant's baseline may indicate progression or need for further safety monitoring.
Change from Baseline in the Best Corrected Visual Acuity (BCVA) Letter Score in the Treated Eye During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in visual clarity (corrected with glasses or contact lenses for refractive errors like nearsightedness, farsightedness, or astigmatism) in the treated eye while participants are receiving and completed oral doxycycline.
  This outcome measures whether visual clarity improves in the treated eye while participants are receiving oral doxycycline.
  BCVA is assessed using a special chart called the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
  The number of letters read correctly is recorded as a letter score, ranging from 0 to 100. An increase in score from the baseline may suggest the treatment is helping improve how well someone sees.
  Trial frames with the lens prescription determined at screening will be used for these assessments.
Change from Baseline in the Best Corrected Visual Acuity (BCVA) Letter Score in the Treated Eye - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in visual clarity (corrected with glasses or contact lenses for refractive errors like nearsightedness, farsightedness, or astigmatism) in the treated eye after participants stop taking oral doxycycline during the long-term follow-up period.
  BCVA is assessed using a special chart called Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
  The number of letters read correctly is recorded as a letter score, ranging from 0 to 100. A drop in score from baseline may indicate a safety issue affecting vision, while stable or improved scores suggest no adverse impact.
  Trial frames with the lens prescription determined at screening will be used for these assessments.
Change from Baseline in Humphrey Visual Field (HVF) Test Results During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in central and peripheral (side) field of vision while participants are receiving and completed oral doxycycline.
  The field of vision is assessed using the Humphrey Visual Field (HVF) test, which checks how well a person can see lights that flash in different areas of their visual field while they focus on a central point.
  Results are reported as a Mean Deviation (MD) score in decibels (dB). For participants with open-angle glaucoma (OAG), the test uses the SITA Standard 24-2 protocol. For participants with non-arteritic anterior ischemic optic neuropathy (NAION), a larger light stimulus (size V) is used.
  Compared to baseline, a more negative MD score means more vision loss, while scores closer to zero suggest better or more normal vision. Improvements in MD from baseline may suggest a positive effect of the treatment.
Change from Baseline in Humphrey Visual Field (HVF) Test Results - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in peripheral (side) field of vision after participants stop taking oral doxycycline during the long-term follow-up period.
  Peripheral field of vision vision is assessed using the Humphrey Visual Field (HVF) test, which checks how well a person can see lights that flash in different areas of their visual field while they focus on a central point.
  Results are reported as a Mean Deviation (MD) score in decibels (dB). For participants with open-angle glaucoma (OAG), the test uses the SITA Standard 24-2 protocol.For participants with non-arteritic anterior ischemic optic neuropathy (NAION), a larger light stimulus (size V) is used.
  A more negative MD score comparing to baseline means more vision loss, and a significant worsening in MD may suggest a safety concern.
Change from Baseline in Quantitative Contrast Sensitivity Function (qCSF) During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in contrast sensitivity while participants are receiving and completed oral doxycycline.
  The quantitative Contrast Sensitivity Function (qCSF), also called quick CSF, is a computerized test that evaluates how well a person can detect differences in contrast - for example, the ability to discern subtle differences in shading or light and dark between an object and its background.
  Higher scores suggest better visual function, while lower scores may indicate difficulty seeing in low-contrast or low-light conditions. Changes in these scores from baseline may reflect signs that the treatment is causing effects.
Change from Baseline in Quantitative Contrast Sensitivity Function (qCSF) - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in contrast sensitivity after participants stop taking oral doxycycline during the long-term follow-up period.
  The quantitative Contrast Sensitivity Function (qCSF), also called quick CSF, is a computerized test that evaluates how well a person can detect differences in contrast - for example, for example, the ability to discern subtle differences in shading or light and dark between an object and its background.
  Lower scores than the baseline values may indicate worsening visual function, and a significant decline in one or more parameters may suggest a safety concern. Changes in these scores from baseline are monitored to see if there are signs that the treatment is causing effects or that the disease is getting worse.
Change from Baseline in Pattern Electroretinogram (pERG) During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in retinal function while participants are receiving and completed oral doxycycline.
  The pERG is a test that checks how well the retina responds to visual patterns like black and white stripes. It helps evaluate the health of retinal ganglion cells, which are important for sending visual signals to the brain.
  The test provides two types of results:
  * Amplitude (measured in microvolts, µV): This shows the strength of the retina's response.
  * Peak time (measured in milliseconds, ms): This shows how quickly the retina responds.
  Higher numbers mean the retina is responding well. Lower numbers or slower response times may suggest that the retina is not working as well as it should. Changes in these results from baseline values may show whether the condition is improving or getting worse during treatment.
Change from Baseline in Pattern Electroretinogram (pERG) - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in retinal function after participants stop taking oral doxycycline during the long-term follow-up period.
  The pERG is a test that checks how well the retina responds to visual patterns like black and white stripes. It helps evaluate the health of retinal ganglion cells, which are important for sending visual signals to the brain.
  The test provides two types of results:
  * Amplitude (measured in microvolts, µV): This shows the strength of the retina's response.
  * Peak time (measured in milliseconds, ms): This shows how quickly the retina responds.
  Lower amplitudes or slower response times than baseline values may indicate worsening retinal function. A significant decline in these results may suggest a safety concern related to signs that the treatment is causing effects or that the disease is getting worse.
Change from Baseline in Optical Coherence Tomography (OCT): Ganglion Cell Layer (GCL) Thickness During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in the thickness of the ganglion cell layer (GCL) while participants are receiving and completed oral doxycycline.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using the Heidelberg Spectralis system.
  The GCL contains the cell bodies of retinal ganglion cells, which are critical for transmitting visual information from the retina to the brain. GCL thickness is measured in micrometers (µm).
  Changes in GCL thickness from baseline values may reflect there are signs that the treatment is causing effects or that the disease is getting worse.
Change from Baseline in Optical Coherence Tomography (OCT): Ganglion Cell Layer (GCL) Thickness - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in the thickness of the ganglion cell layer (GCL) after participants stop taking oral doxycycline during the long-term follow-up period.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using the Heidelberg Spectralis system.
  The GCL contains the cell bodies of retinal ganglion cells, which are critical for transmitting visual information from the retina to the brain. GCL thickness is measured in micrometers (µm).
  A significant decrease in GCL thickness from baseline values may suggest a safety concern related to signs that the treatment is causing effects or that the disease is getting worse.
Change from Baseline in Optical Coherence Tomography (OCT): Retinal Nerve Fiber Layer (RNFL) Thickness During and Post-Doxycycline Activation Period - Efficacy | Baseline to Day 56, Day 112
  This outcome measures the change in the thickness of the retinal nerve fiber layer (RNFL) while participants are receiving and completed oral doxycycline.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using the Heidelberg Spectralis system.
  The RNFL contains nerve fibers that help carry visual signals from the eye to the brain. RNFL thickness is measured in micrometers (µm).
  Changes in RNFL thickness from baseline values may reflect signs that the treatment is causing effects or that the disease is getting worse.
Change from Baseline in Optical Coherence Tomography (OCT): Retinal Nerve Fiber Layer (RNFL) Thickness - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures the change in the thickness of the retinal nerve fiber layer (RNFL) after participants stop taking oral doxycycline during the long-term follow-up period.
  Optical Coherence Tomography (OCT) is a non-invasive imaging test that uses light waves to take detailed cross-sectional pictures of the retina. OCT will be conducted using the Heidelberg Spectralis system.
  The RNFL contains nerve fibers that help carry visual signals from the eye to the brain. RNFL thickness is measured in micrometers (µm).
  A significant decrease in RNFL thickness from baseline values may suggest a safety concern related to signs that the treatment is causing effects or that the disease is getting worse.
Change in Neutralizing Antibodies (NAbs) to AAV2 During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This outcome measures changes in the body's immune response to the AAV2 virus while participants are receiving and completed oral doxycycline.
  Specifically, it looks at neutralizing antibodies, which are proteins made by the immune system that can block the virus from working.
  Blood samples are tested to see how much antibody is present. The results are reported as a number called a "titer," which shows how strong the response is.
  * A higher titer means the body is making more antibodies that can block the virus.
  * A lower titer or no detectable antibodies means the virus is less likely to be blocked.
  These results help researchers understand how the body reacts to the treatment and whether the immune system might affect how well the therapy works.
Change in Cellular Immune Response to ER-100 Peptides via ELISpot During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This outcome measures how the immune system's T cells respond to parts of the ER-100 treatment while participants are receiving and completed oral doxycycline.
  A lab test called ELISpot is used to count how many immune cells release a signal when they recognize parts of the treatment.
  Each signal shows up as a spot in the test - more spots mean a stronger immune response, and fewer spots mean a weaker response.
  This helps researchers understand how active the immune system is and whether it might affect how well the treatment works or how the body tolerates it.
Change in ER-100 Viral Shedding via qPCR to During and Post-Doxycycline Activation Period | Baseline to Day 56, Day 112
  This outcome measures whether any part of the ER-100 treatment is released from the body while participants are receiving and completed oral doxycycline.
  Samples are collected from tears, nasal swab, saliva, blood, urine, and feces. A lab test called qPCR is used to detect tiny amounts of ER-100 DNA in these fluids.
  If ER-100 DNA is found, it means the treatment is leaving the body through these fluids - this is called viral shedding.
  If no ER-100 DNA is found, it means the treatment is staying inside the body. More shedding may suggest the body is clearing the treatment faster, while less or no shedding may mean the treatment is staying localized or being retained longer.
  This helps researchers understand how the treatment moves through the body and whether it could be passed to others.
Change in Biodistribution of ER-100 Vector DNA in Aqueous Humor During Doxycycline Activation Period | Baseline to Day 56
  This outcome measures whether any part of the ER-100 treatment is found in the fluid inside the eye (called aqueous humor) while participants are receiving oral doxycycline.
  This test is only done in participants with open-angle glaucoma (OAG).
  A lab test called qPCR is used to detect tiny amounts of ER-100 DNA in the eye fluid.
  * If ER-100 DNA is found, it means the treatment has reached the inside of the eye.
  * If no ER-100 DNA is found, it means the treatment has not entered that part of the eye.
  This helps researchers understand where the treatment travels in the body and whether it stays in the intended area.
Change from Baseline in Slit Lamp Exam Results - Long-term Follow-up Period - Safety | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures changes in the health of the front structures of the eye after participants stop taking oral doxycycline during the long-term follow-up period.
  A slit lamp exam is a routine eye test that uses a bright light and microscope to closely examine the front parts of the eye, including the cornea, iris, lens, and the white part of the eye. The exam helps detect signs of irritation, inflammation, infection, or other damage.
  Changes from baseline observed during the slit lamp exam might be signs that the treatment is causing effects or that the disease is getting worse.
Incidence of Treatment-Emergent Adverse Events (TEAEs) - Long-term Follow-up Period | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome tracks any new or worsening health problems that occur after participants stop taking oral doxycycline during the long-term follow-up period.
  These health problems are called treatment-emergent adverse events (TEAEs). Researchers record how often these events happen, what kind they are (such as headaches, infections, or changes in lab tests), and how serious they are.
  This helps determine whether the ER-100 treatment causes any long-term side effects or health concerns, even months or years after the initial treatment.
Change in Safety Laboratory Test Results - Long-term Follow-up Period | Baseline to Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  This outcome measures changes in routine lab test results after participants stop taking oral doxycycline, during the long-term follow-up period.
  These tests check things like liver and kidney function, blood counts, and other indicators of general health.
  If lab values change over time, it may show how the body is responding to the ER-100 treatment in the long term.
  This helps researchers monitor for any delayed side effects or health concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Rosenzweign-Lipson, PhD, Study Chair — Life Biosciences Inc.
Locations (1):
- Global Research Management, Inc., Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not yet been finalized. Data sharing may be considered after study completion, depending on regulatory guidance, publication requirements, and available resources to support secure access.